CLINICAL TRIAL: NCT03766984
Title: Study of Non-pharmacokinetic Interaction Between Diclofenac 25 mg and 25 mg Tramadol With the Fixed-dose Combination Tablets of the Two Drugs Administered to Healthy Subjects of Both Genders in Fasting State
Brief Title: Pharmacokinetic Non-interaction Study With a Fixed-dose Combination Tablet With Tramadol and Diclofenac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Grünenthal Colombiana S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DCLF/TRMD-GRNN-01; HP8001-01 (Other: Grünenthal)
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Pharmacokinetics
Keywords: fixed-dose combination; diclofenac; tramadol; interaction
MeSH Terms: interventions — Diclofenac; Tramadol

STUDY DESIGN:
Intervention Model Description: Longitudinal, prospective, crossover, open, randomized, single-dose study with 3 periods, 2 sequences (ACB and BCA), and 3 treatments (A, B, and C) in healthy participants and under fasting conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diclofenac 25 mg (Experimental): Participants receive 1 tablet of diclofenac sodium 25 mg with 250 milliliters of purified water.
  Interventions: Drug: Diclofenac sodium 25 mg
- Tramadol 25 mg (Experimental): Participants receive 1 tablet of tramadol hydrochloride 25 mg with 250 milliliters of purified water.
  Interventions: Drug: Tramadol hydrochloride 25 mg
- Diclofenac/Tramadol 25 mg/25 mg FDC (Experimental): Participants receive 1 fixed-dose combination tablet of diclofenac sodium 25 mg/tramadol hydrochloride 25 mg with 250 milliliters of purified water.
  Interventions: Drug: Diclofenac sodium 25 mg/Tramadol hydrochloride 25 mg

INTERVENTIONS:
Drug: Diclofenac sodium 25 mg — Diclofenac sodium 25 mg Tablets (Laboratorios Tecnandina S.A., Ecuador)
  Arms: Diclofenac 25 mg
Drug: Tramadol hydrochloride 25 mg — Tramadol hydrochloride 25 mg Tablets (Laboratorios Tecnandina S.A., Ecuador)
  Arms: Tramadol 25 mg
Drug: Diclofenac sodium 25 mg/Tramadol hydrochloride 25 mg — Fixed-dose combination tablet containing diclofenac sodium 25 mg and tramadol hydrochloride 25 mg (Laboratorios Tecnandina S.A., Ecuador)
  Other Names: Adorlan (Trade Mark)
  Arms: Diclofenac/Tramadol 25 mg/25 mg FDC

SUMMARY:
The objective of the study was to evaluate whether or not there is a substantial pharmacokinetic interaction between diclofenac and tramadol in a new formulation of a fixed-dose combination of diclofenac 25 milligrams (mg) and tramadol 25 mg for oral administration. The study was conducted in healthy participants of both genders.

DETAILED DESCRIPTION:
After a screening period of about 2 weeks, 36 eligible healthy men and women were randomly allocated to receive 3 sequential treatments in the following order:

* a single dose of diclofenac followed by a single dose of the fixed-dose combination of diclofenac/tramadol followed by a single dose of tramadol
* a single dose of tramadol followed by a single dose of the fixed-dose combination of diclofenac/tramadol followed by a single dose of diclofenac.

There were washout periods of 7 days between treatments.

Sixteen blood samples were collected per participant: at pre-dose and 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 and 36 hours after administration of each of the study drugs.

The pharmacokinetic parameters and relative bioavailabilities of diclofenac and tramadol (and of the tramadol metabolite M1) were determined for the new fixed-dose combination product and were compared to the single compound reference products.

Furthermore, the safety (frequency of adverse events) and tolerability of the new fixed-dose combination of diclofenac 25 mg and 25 mg tramadol in healthy men and women was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 and 55 years of age.
* Women with use of a barrier method as a contraceptive.
* Body mass index equal to or above 18.0 and equal to or less than 27.0 kilograms per square meter.
* Clinically healthy. If the clinical history, the registration of vital signs and the physical examination did not show abnormal deviations that avoid their participation in a clinical study.
* Without a history of allergic reactions to the study drug.
* Stable vital signs during the selection (heart rate, respiratory rate, blood pressure at rest and axillary body temperature).
* Laboratory studies: complete blood count, blood chemistry of 24 items, urinalysis, anti-human immunodeficiency virus (HIV) 1, anti-HIV2, anti-hepatitis B surface antigen (HBs) and anti-hepatitis C virus (HCVs) antibodies, and serologic test for syphilis [Venereal Disease Research Laboratory test]) within normal ranges according to the reference laboratory, or that the deviations are not clinically significant. If the deviation has no clinical significance, it may be justified the inclusion of the participant to the clinical study. The age of the report of the clinical laboratory studies must not be greater than 3 months.
* Electrocardiogram (ECG) with no pathological alterations, with validity of no more than 3 months.
* The participant accepts the restrictions and indications described in the protocol and internal regulations.
* The participant has read and understood the relevant aspects of the clinical study and gives its authorization for participation by signing the informed consent form before inclusion on the clinical study and performing any procedure.

Exclusion Criteria:

* Findings in the clinical history, vital signs and/or physical examination that show abnormal conditions of the general state of health of the participant that avoid its participation in a clinical study.
* Recent exposure to the study drug between the 30 days prior or any other medication by prescription or self consumed between the 14 days prior to the start of the study, or that do not accept to avoid its consumption during the course of the study.
* Surgery during the 30 days prior to the start of the study.
* Suspicion or evidence of infection by Human Immunodeficiency Virus (HIV), hepatitis B virus (HBV) and/or hepatitis C virus (HCV).
* Serologic test for syphilis (Venereal Disease Research Laboratory test) positive.
* Known hypersensitivity to any medication.
* Blood donation equal to or above 1 unit (0.5 liters) during the 30 days prior to the selection.
* Participants who have special food requirements or food restrictions.
* Women in the breastfeeding period and/or pregnant.
* Positive results in the qualitative test of pregnancy in urine (only women).
* Positive result in the qualitative detection of drugs of abuse.
* Participation in a clinical study Phase 1, 2 or 3 or bioavailability/ bioequivalence studies during the 3 months previous to the selection.
* The participant does not give his or her authorization to participate in the study through the signing of an informed consent, or is not willing to follow the indications and/or restrictions of the protocol and rules of the procedure.
* The participant is vulnerable or potentially vulnerable by which cannot freely express his/her consent by subordination of the principal investigator or by coercion of any third party.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-06-07 (Actual); Primary Completion 2015-06-23 (Actual); Study Completion 2015-06-23 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of diclofenac | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Diclofenac concentrations were determined using validated analytical methods.
Maximum plasma concentration (Cmax) of tramadol | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Tramadol concentrations were determined using validated analytical methods.
Area under the plasma concentration curve from the administration until the time t (AUC0-t) of diclofenac | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Diclofenac concentrations were determined using validated analytical methods.
Area under the plasma concentration curve from the administration until the time t (AUC0-t) of tramadol | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Tramadol concentrations were determined using validated analytical methods.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of tramadol metabolite M1 | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Tramadol M1 concentrations were determined using validated analytical methods.
Area under the plasma concentration curve from the administration until the time t (AUC0-t) of tramadol metabolite M1 | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Tramadol M1 concentrations were determined using validated analytical methods.
Area under the plasma concentration curve from 0 to infinity (AUC0-inf) of tramadol | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Tramadol concentrations were determined using validated analytical methods.
Area under the plasma concentration curve from 0 to infinity (AUC0-inf) of tramadol metabolite M1 | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Tramadol M1 concentrations were determined using validated analytical methods.
Area under the plasma concentration curve from 0 to infinity (AUC0-inf) of diclofenac | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Diclofenac concentrations were determined using validated analytical methods.
Time to maximum plasma concentration (Tmax) for tramadol | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Tmax was calculated based on Cmax data for tramadol.
Time to maximum plasma concentration (Tmax) for tramadol metabolite M1 | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Tmax was calculated based on Cmax data for tramadol M1.
Time to maximum plasma concentration (Tmax) for diclofenac | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. Tmax was calculated based on Cmax data for diclofenac
Elimination half life (t half) for tramadol | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. t half was calculated based on plasma concentration data for tramadol.
Elimination half life (t half) for tramadol metabolite M1 | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. T half was calculated based on plasma concentration data for tramadol M1.
Elimination half life (t half) for diclofenac | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. t half was calculated based on plasma concentration data for diclofenac.
Elimination rate constant (KE) for tramadol | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. KE will be calculated based on the plasma concentrations for tramadol.
Elimination rate constant (KE) for tramadol metabolite M1 | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. KE was calculated based on the plasma concentrations for tramadol M1.
Elimination rate constant (KE) for diclofenac | From pre-dose to 36 hours post-dose
  16 plasma samples were collected from pre-dose to 36 hours post-dose. KE will be calculated based on the plasma concentrations for diclofenac.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Clinical Unit of Biodextra, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Web Site (see URL below for details)
Supporting Information: Study Protocol, SAP, CSR
URL: http://www.grunenthal.com/r-d-vision-mission/clinical-trials/data-sharing-clinical-trials